CLINICAL TRIAL: NCT07260123
Title: Medicolegal Aspects of Traumatic Hand Injuries in the Period From October 2025 to April 2026 in Sohag University Hospitals
Brief Title: Medicolegal Aspects of Traumatic Hand Injuries
Acronym: hand-injuries
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Abdellah Ahmed, Demonstrator of Forensic Medicine & Clinical Toxicology Faculty of Medicine Sohag University, Sohag University
Other Study IDs: Soh-Med-25-9---21MS
Record Dates: First submitted 2025-09-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Hand Injuries; Medicolegal Aspects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosed cases with traumatic hand and wrist injuries: Diagnosed cases with traumatic hand and wrist injuries of any age ,sex, educational level

SUMMARY:
The goal of this observational study is to assess and describe the epidemiology of traumatic hand injuries in Sohag University Hospital in different age group ,male, female with traumatic hand injury The main questions it aims to answer are:

what is the mechanism of injury ? what is the outcome of the injury ?

DETAILED DESCRIPTION:
The goal of this observational study is to assess and describe the epidemiology of traumatic hand injuries in Sohag University Hospital. study and analyze the medicolegal aspects of different traumatic hand injuries cases (patterns of injuries, mechanisms, causes, site of trauma and outcomes) in different age group ,male, female with traumatic hand injury The main questions it aims to answer are:

what is the mechanism of injury ? what is the Manner of Injury ? what is the outcome of the injury ? hs the injury affect the function of the hand ?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases with traumatic hand and wrist injuries
* Patient is willing to attend follow up appointments

Exclusion Criteria:

* Patients with deficient data i.e. escaped, discharged on demand before period of follow up,…etc
* Patient presented by life threating injuries in addition to hand injuries.
* Patient with previous pathology in hand.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is specified in sohag university hospitals on patients with traumatic hand injuries
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
assess the incidance of traumatic hand injuries in Sohag University Hospital in a period from October 2025 to April 2026 | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No